CLINICAL TRIAL: NCT03253796
Title: A Phase-IV, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Evaluate the Efficacy and Safety of Golimumab (MK-8259 [SCH 900259]) After Treatment Withdrawal, Compared With Continued Treatment (Either Full- or Reduced-Treatment Regimen), In Subjects With Non-Radiographic Axial Spondyloarthritis
Brief Title: Golimumab (MK-8259 / SCH900259) Treatment Withdrawal in Participants With Non-radiographic Axial Spondyloarthritis (GO-BACK) (MK-8259-038)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8259-038; MK-8259-038 (Other: Merck); 2015-004020-65 (EudraCT Number)
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — golimumab

STUDY DESIGN:
Intervention Model Description: To evaluate the effect of treatment withdrawal compared to continued treatment with golimumab (either every month [QM] or every 2 months [Q2M]) on the incidence of a "flare" during up to 12 months in Period 2 (blinded therapy).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GLM SC QM (Full Treatment Regimen) (Experimental): Period 1: participants are treated with open-label (OL) GLM SC QM for up to 10 months; Period 2: participants are treated with double-blinded SC GLM QM for up to 12 months
  Interventions: Biological: Golimumab
- GLM SC Q2M (Reduced Treatment Regimen) (Experimental): Period 1: participants are treated with OL GLM SC QM for up to 10 months; Period 2: participants are treated with double-blinded GLM SC every other month alternating with matching placebo to GLM every other month for up to 12 months
  Interventions: Biological: Golimumab; Biological: Placebo
- Placebo (Treatment Withdrawal Regimen) (Placebo Comparator): Period 1: participants are treated with OL GLM SC QM for up to 10 months; Period 2: participants are treated with double-blinded placebo for up to 12 months
  Interventions: Biological: Golimumab; Biological: Placebo
- OL GLM Retreatment (Experimental): Participants who experience a disease flare during double-blinded treatment in Period 2 will discontinue blinded treatment and receive OL GLM SC QM.
  Interventions: Biological: Golimumab

INTERVENTIONS:
Biological: Golimumab — Injections of 50 mg golimumab. At the investigator's discretion, participants with a body weight of more than 100 kg could receive 100 mg injections with golimumab.
  Other Names: MK-8259; Simponi®
Biological: Placebo — Injections of matching placebo for golimumab.
  Arms: GLM SC Q2M (Reduced Treatment Regimen); Placebo (Treatment Withdrawal Regimen)

SUMMARY:
The purpose of this study is to evaluate the effect of treatment withdrawal compared to continued treatment with golimumab (GLM) administered by subcutaneous (SC) injection on the incidence of a "flare" in non-radiographic axial spondyloarthritis over up to 12 months. The primary hypothesis is that continued treatment with golimumab is superior to treatment withdrawal, based on the percentage of subjects without a "flare" during up to 12 months of blinded therapy.

ELIGIBILITY:
Inclusion Criteria:

* Is not of reproductive potential, or is of reproductive potential and agrees to avoid becoming pregnant or impregnating a partner while receiving trial medication or within 6 months after the last dose of trial medication
* Has chronic back pain of ≥3 months duration by history
* Has physician-diagnosed active non-radiographic axial spondyloarthritis (nr-axSpA) with disease duration <= 5 years
* Meets one of the following criteria:

  1. Has active inflammation on magnetic resonance imaging (MRI) highly suggestive of sacroiliitis associated with spondyloarthropathy and 1 or more of the following spondyloarthritis (SpA) characteristics:

     * Inflammatory back pain
     * Arthritis (physician-diagnosed)
     * Enthesitis (heel) physician-diagnosed (spontaneous pain or tenderness at examination of the site of the insertion of the Achilles tendon or plantar fascia)
     * Dactylitis (physician-diagnosed)
     * Psoriasis (physician-diagnosed)
     * History of physician-diagnosed inflammatory bowel disease (IBD)
     * History of uveitis confirmed by an ophthalmologist
     * Good response to nonsteroidal anti-inflammatory drugs (NSAID)
     * Family history of SpA (presence of ankylosing spondylitis, psoriasis, acute uveitis, reactive arthritis, or IBD)
     * Elevated C-reactive protein (CRP)

       * Human leukocyte antigen B27 (HLA-B27)+ gene OR
  2. Has a HLA-B27+ gene and 2 or more of the following SpA characteristics:

     * Inflammatory back pain
     * Arthritis (physician-diagnosed)
     * Enthesitis (heel) physician-diagnosed (spontaneous pain or tenderness at examination of the site of the insertion of the Achilles tendon or plantar fascia)
     * Dactylitis (physician-diagnosed)
     * Psoriasis (physician-diagnosed)
     * History of physician-diagnosed inflammatory bowel disease (IBD)
     * History of uveitis confirmed by an ophthalmologist
     * Good response to nonsteroidal anti-inflammatory drugs (NSAID)
     * Family history of SpA (presence of ankylosing spondylitis, psoriasis, acute uveitis, reactive arthritis, or IBD)
     * Elevated C-reactive protein (CRP)
* Has elevated CRP at Screening or evidence of active inflammation in the sacroiliac joints on MRI
* Has an Ankylosing Spondylitis Disease Activity Score (ASDAS) >= 2.1 at Screening
* Shows high disease activity at Screening and Baseline of both a Total Back Pain score of ≥4 and a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of >= 4
* Has an acceptable history of NSAID use
* Has no history of untreated latent or active tuberculosis (TB) prior to Screening
* Has had no recent close contact with a person with active TB or, if there has been such contact, will undergo additional evaluations and receive appropriate treatment for latent TB
* Agrees to undergo screening for hepatitis B virus (HBV) and demonstrates negative results for hepatitis B surface antigen (HBsAg) and HBV deoxyribonucleic acid (DNA)

Exclusion Criteria:

* Has bilateral sacroiliitis Grade 2 or unilateral sacroiliitis Grade 3 or Grade 4 on conventional x-rays
* Is a nursing or pregnant female, or intends to become pregnant within 6 months after receiving trial medication
* Intends to donate eggs (female participants) or sperm (male participants) while receiving trial medication or within 6 months after trial medication
* Has any clinically significant condition or situation that would interfere with the trial evaluations or participation in the trial
* Has ever received any cytotoxic drugs, including chlorambucil, cyclophosphamide, nitrogen mustard, or other alkylating agents
* Has received any treatment listed below more recently than the indicated off-drug period prior to Screening

  * • Disease-modifying anti-rheumatic drugs (30 days off drug)
  * • Live vaccinations (3 months off drug)
  * • Investigational medications (30 days or 5 half-lives off drug, whichever is longer)
  * • Bacille Calmette-Guerin (BCG) vaccination (12 months off drug)
* Has any systemic inflammatory condition, including psoriatic arthritis, active Lyme disease, systemic lupus erythematosus, infectious arthritis, vasculitis, parvovirus infection, rheumatoid arthritis, active uveitis, or active IBD
* Has a history of latent or active granulomatous infection prior to Screening
* Had a nontuberculous mycobacterial infection or opportunistic infection within 6 months prior to Screening
* Has a history of an infected joint prosthesis, or has received antibiotics for a suspected infection of a joint prosthesis, if that prosthesis has not been removed or replaced
* Had a serious infection, has been hospitalized for an infection, or has been treated with IV antibiotics for an infection within 2 months prior to Baseline
* Had a history of, or ongoing, chronic or recurrent infectious disease
* Is known to be infected with human immunodeficiency virus (HIV) or seropositive for hepatitis C virus (HCV)
* Has had a chest x-ray within 2 months prior to Screening that shows an abnormality suggestive of a current active infection or malignancy
* Has a history of lymphoproliferative disease
* Has had a malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of cervix that has been surgically cured)
* Has a history of known demyelinating diseases such as multiple sclerosis or optic neuritis
* Has a history of or concurrent congestive heart failure of any grade
* Has a transplanted organ (with the exception of a corneal transplant performed >= 3 months prior to baseline)
* Has current signs or symptoms of significant medical illness which could interfere with the trial, or require treatment that might interfere with the trial
* Is a user of recreational or illicit drugs or has or had a substance abuse (drug or alcohol) problem within the previous 2 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (71):
- Czechia (9):
  - FN Brno ( Site 0005), Brno
  - Revmatologie s.r.o. ( Site 0009), Brno
  - CCBR Ostrava s.r.o. ( Site 0001), Ostrava
  - Artroscan s.r.o. ( Site 0007), Ostrava-Trebovice
  - CCR Czech a.s. ( Site 0003), Pardubice
  - CCR Prague s.r.o ( Site 0004), Prague
  - Fakultni nemocnice v Motole ( Site 0127), Prague
  - Medical Plus s.r.o ( Site 0010), Uherské Hradiště
  - PV - Medical s.r.o. ( Site 0006), Zlín
- Germany (5):
  - Universitaetsklinik der Charite Berlin ( Site 0023), Berlin
  - U. klinikum Koeln AOER ( Site 0025), Cologne
  - Rheumazentrum Ruhrgebiet ( Site 0021), Herne
  - Klinikum der Universitaet Muenchen - LMU ( Site 0026), München
  - Herbert Kellner Innere Medizin Rheumatologie und Gastroenterologie ( Site 0022), München
- Netherlands (4):
  - Antonius Ziekenhuis Sneek ( Site 0043), Sneek, Provincie Friesland
  - Vrij Universiteit Medisch Centrum ( Site 0044), Amsterdam
  - Leids Universitair Medisch Centrum ( Site 0041), Leiden
  - Maasstad Ziekenhuis ( Site 0042), Rotterdam
- Poland (11):
  - Prywatna Praktyka Lekarska, Dr. med. Pawel Hrycaj ( Site 0060), Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Katowice ( Site 0059), Katowice, Silesian Voivodeship
  - NZOZ Osteo-Medic s.c. A. Racewicz, R. Supronik ( Site 0058), Bialystok
  - Klinika Reumatologii i Ukladowych Chorob Tkanki Lacznej ( Site 0153), Bydgoszcz
  - Centrum Kliniczno-Badawcze ( Site 0152), Elblag
  - Krakow Medical Centre ( Site 0052), Krakow
  - NZOZ Reumed ( Site 0051), Lublin
  - Pomorskie Cent. Reumatologiczne IM.Dr. Titz-Kosko W Sopocie Sp. Z.o.o. ( Site 0057), Sopot
  - Lubelskie Centrum Diagnostyczne ( Site 0053), Świdnik
  - NZOZ Nasz Lekarz Praktyka Grupowa Lekarzy Rodzinnych ( Site 0151), Torun
  - Reumatika ( Site 0055), Warsaw
- Romania (10):
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed ( Site 0177), Brasov
  - Clinical Hospital Ioan Cantacuzino ( Site 0184), Bucaresti
  - SC Duo Medical SRL ( Site 0183), Bucharest
  - Spitalul Clinic Sfanta Maria ( Site 0182), Bucharest
  - Colentina Clinical Hospital ( Site 0231), Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca ( Site 0176), Cluj-Napoca
  - RKMed Center ( Site 0180), Iași
  - S.C.Pelican Impex S.R.L ( Site 0232), Oradea
  - Covamed Serv SRL ( Site 0178), Sfântu Gheorghe
  - Cabinet Medical Medicina Interna Dr. Triff Carina ( Site 0179), Timișoara
- Russia (7):
  - GUZ Regional Clinical Hospital ( Site 0076), Saratov, Oktyabrskiy Region
  - Rheumatology Research Institute n.a. V.A.Nasonova of RAMS ( Site 0061), Moscow
  - SPb SBHI Clinical Rheumatological Hospital 25 ( Site 0077), Saint Petersburg
  - SBHI Leningrad Regional Clinical Hospital ( Site 0065), Saint Petersburg
  - LLC Sanavita ( Site 0074), Saint Petersburg
  - Tolyatti City Clinical Hospital 5 ( Site 0069), Tolyatti
  - Yaroslavl Clinical Hospital for Emergency Care na. NV. Solovyev. ( Site 0075), Yaroslavl
- Spain (4):
  - Hospital de Basurto ( Site 0082), Bilbao
  - Hospital Universitario Reina Sofia ( Site 0081), Córdoba
  - Hospital Universitario La Paz ( Site 0083), Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca ( Site 0085), Murcia
- Turkey (Türkiye) (7):
  - Akdeniz Universitesi Tip Fakultesi Romatoloji Departmani ( Site 0094), Antalya, Ankara
  - Ankara Numune Egitim Arastirma Hastanesi ( Site 0092), Ankara
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 0091), Ankara
  - Ankara Universitesi Tıp Fakultesi ( Site 0093), Ankara
  - Pamukkale Unv. Tip Fak. ( Site 0097), Denizli
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 0098), Istanbul
  - Kocaeli Universitesi Tip Fakultesi Ic Hastaliklari ( Site 0096), Kocaeli
- Ukraine (14):
  - Cherkassy Regional hospital of Cherkassy Regional council ( Site 0221), Cherkassy
  - MI Dnipr Regional Clinical Hospital named after I.I. Mechnikov ( Site 0222), Dnipropetrovsk
  - SI National Institute of therapy n.a L.T. Maloi NAMS of Ukraine ( Site 0261), Kharkiv
  - ME of Health Care Kharkiv City Clinical Hospital #8 ( Site 0262), Kharkiv
  - Kyivska miska klinichna likarnia N3 ( Site 0266), Kyiv
  - M. D. Strazhesko Institute of Cardiology. ( Site 0264), Kyiv
  - Medical Center Ibn Sina ( Site 0268), Kyiv
  - Clinic of Modern Rheumatology ( Site 0265), Kyiv
  - Communal City Clinical Hospital #4 ( Site 0230), Lviv
  - MI Odesa Regional Clinical Hospital ( Site 0226), Odesa
  - M.V.Sklifosovskyi Poltava Regional Clinical Hospital ( Site 0224), Poltava
  - Vinnitsa Regional Clinical Hospital n.a. Pirogov ( Site 0225), Vinnutsya
  - SRI of Invalid Rehabilitation of Vinnytsia M.I.Pyrogov ( Site 0263), Vinnytsia
  - Zaporizhzha Regional Clinical Hospital ( Site 0223), Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Weinstein CLJ, Sliwinska-Stanczyk P, Hala T, Stanislav M, Tzontcheva A, Yao R, Berd Y, Curtis SP, Philip G. Efficacy and safety of golimumab in patients with non-radiographic axial spondyloarthritis: a withdrawal and retreatment study (GO-BACK). Rheumatology (Oxford). 2023 Nov 2;62(11):3601-3609. doi: 10.1093/rheumatology/kead112. PMID 36919768

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Run-In Golimumab QM: Participants were treated with open-label subcutaneous (SC) injections of 50 mg golimumab once a month (QM) for up to 10 months. Participants with a body weight greater than 100 kg may have received 100 mg injections of golimumab at the discretion of the investigator.
- Golimumab QM (Full Treatment Regimen): Participants were treated with double-blinded SC injections of 50 mg golimumab QM for up to 12 months. Participants with a body weight greater than 100 kg who had received 100 mg injections of golimumab in Period 1 continued to receive this dosage for the duration of the study. Participants who experienced a disease flare during double-blinded treatment in Period 2 discontinued blinded treatment and were retreated with open-label golimumab.
- Golimumab Q2M (Reduced Treatment Regimen): Participants were treated with double-blinded SC injections of 50 mg golimumab every other month (Q2M) alternating with matching placebo to golimumab every other month for up to 12 months. Participants with a body weight greater than 100 kg who had received 100 mg injections of golimumab in Period 1 continued to receive this dosage for the duration of the study. Participants who experienced a disease flare during double-blinded treatment in Period 2 discontinued blinded treatment and were retreated with open-label golimumab.
- Placebo (Treatment Withdrawal Regimen): Participants were treated with double-blinded SC injections of placebo for up to 12 months. Participants who experienced a disease flare during double-blinded treatment in Period 2 discontinued blinded treatment and were retreated with open-label golimumab.
- Open-Label Retreatment: Participants who experienced a disease flare were treated with open-label SC injections of 50 mg golimumab QM for up to 12 months. Participants with a body weight greater than 100 kg who had received 100 mg injections of golimumab in Period 1 continued to receive this dosage for the duration of the study.
Period: Period 1: Run-In
Arm/Group | Open-Label Run-In Golimumab QM | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment
Started | 323 | 0 | 0 | 0 | 0
Completed | 207 | 0 | 0 | 0 | 0
Not Completed | 116 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Qualifying Event | 98 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0 | 0 | 0
Period: Period 2: Withdrawal vs Continued Tx
Arm/Group | Open-Label Run-In Golimumab QM | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment
Started (18 participants did not continue into Period 2) | 0 | 63 | 64 | 62 | 0
Completed | 0 | 53 | 43 | 21 | 0
Not Completed | 0 | 10 | 21 | 41 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3 | 0
Not completed — Did not attain inactive disease in Period 1 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Flare, transitioned to Open-label retreatment | 0 | 10 | 15 | 38 | 0
Period: Period 2: Open-Label Retreatment
Arm/Group | Open-Label Run-In Golimumab QM | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment
Started | 0 | 0 | 0 | 0 | 63
Completed | 0 | 0 | 0 | 0 | 58
Not Completed | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-Label Run-In Golimumab QM | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment | Total
Number analyzed (Participants) | 323 | 63 | 64 | 62 | 63 | 575
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The first row represents Period 1, the second row represents the double-blind portion of Period 2, and the third row represents open-label retreatment in Period 2
  Years
    Period 1: Open-Label Run-In: number analyzed (Participants) | 323 | 0 | 0 | 0 | 0 | 323
    Period 1: Open-Label Run-In | 32.5 (7.2) |  |  |  |  | 32.5 (7.2)
    Period 2: Withdrawal vs Continued Tx: number analyzed (Participants) | 0 | 63 | 64 | 62 | 0 | 189
    Period 2: Withdrawal vs Continued Tx |  | 31.4 (8.0) | 30.8 (6.7) | 32.9 (6.8) |  | 31.7 (7.2)
    Period 2: Open-Label Retreatment: number analyzed (Participants) | 0 | 0 | 0 | 0 | 63 | 63
    Period 2: Open-Label Retreatment |  |  |  |  | 33.4 (6.7) | 33.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The first row represents Period 1, the second row represents the double-blind portion of Period 2, and the third row represents open-label retreatment in Period 2
  Participants
    Period 1: Open-Label Run-In: number analyzed (Participants) | 323 | 0 | 0 | 0 | 0 | 323
    Period 1: Open-Label Run-In: Female | 109 |  |  |  |  | 109
    Period 1: Open-Label Run-In: Male | 214 |  |  |  |  | 214
    Period 2: Withdrawal vs Continued Tx: number analyzed (Participants) | 0 | 63 | 64 | 62 | 0 | 189
    Period 2: Withdrawal vs Continued Tx: Female |  | 19 | 21 | 16 |  | 56
    Period 2: Withdrawal vs Continued Tx: Male |  | 44 | 43 | 46 |  | 133
    Period 2: Open-Label Retreatment: number analyzed (Participants) | 0 | 0 | 0 | 0 | 63 | 63
    Period 2: Open-Label Retreatment: Female |  |  |  |  | 20 | 20
    Period 2: Open-Label Retreatment: Male |  |  |  |  | 43 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The first row represents Period 1, the second row represents the double-blind portion of Period 2, and the third row represents open-label retreatment in Period 2
  Participants
    Period 1: Open-Label Run-In: number analyzed (Participants) | 323 | 0 | 0 | 0 | 0 | 323
    Period 1: Open-Label Run-In: Hispanic or Latino | 2 |  |  |  |  | 2
    Period 1: Open-Label Run-In: Not Hispanic or Latino | 321 |  |  |  |  | 321
    Period 1: Open-Label Run-In: Unknown or Not Reported | 0 |  |  |  |  | 0
    Period 2: Withdrawal vs Continued Tx: number analyzed (Participants) | 0 | 63 | 64 | 62 | 0 | 189
    Period 2: Withdrawal vs Continued Tx: Hispanic or Latino |  | 0 | 0 | 0 |  | 0
    Period 2: Withdrawal vs Continued Tx: Not Hispanic or Latino |  | 63 | 64 | 62 |  | 189
    Period 2: Withdrawal vs Continued Tx: Unknown or Not Reported |  | 0 | 0 | 0 |  | 0
    Period 2: Open-Label Retreatment: number analyzed (Participants) | 0 | 0 | 0 | 0 | 63 | 63
    Period 2: Open-Label Retreatment: Hispanic or Latino |  |  |  |  | 0 | 0
    Period 2: Open-Label Retreatment: Not Hispanic or Latino |  |  |  |  | 63 | 63
    Period 2: Open-Label Retreatment: Unknown or Not Reported |  |  |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The first row represents Period 1, the second row represents the double-blind portion of Period 2, and the third row represents open-label retreatment in Period 2
  Participants
    Period 1: Open-Label Run-In: number analyzed (Participants) | 323 | 0 | 0 | 0 | 0 | 323
    Period 1: Open-Label Run-In: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Period 1: Open-Label Run-In: Asian | 0 |  |  |  |  | 0
    Period 1: Open-Label Run-In: Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  | 0
    Period 1: Open-Label Run-In: Black or African American | 0 |  |  |  |  | 0
    Period 1: Open-Label Run-In: White | 323 |  |  |  |  | 323
    Period 1: Open-Label Run-In: More than one race | 0 |  |  |  |  | 0
    Period 1: Open-Label Run-In: Unknown or Not Reported | 0 |  |  |  |  | 0
    Period 2: Withdrawal vs Continued Tx: number analyzed (Participants) | 0 | 63 | 64 | 62 | 0 | 189
    Period 2: Withdrawal vs Continued Tx: American Indian or Alaska Native |  | 0 | 0 | 0 |  | 0
    Period 2: Withdrawal vs Continued Tx: Asian |  | 0 | 0 | 0 |  | 0
    Period 2: Withdrawal vs Continued Tx: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 |  | 0
    Period 2: Withdrawal vs Continued Tx: Black or African American |  | 0 | 0 | 0 |  | 0
    Period 2: Withdrawal vs Continued Tx: White |  | 63 | 64 | 62 |  | 189
    Period 2: Withdrawal vs Continued Tx: More than one race |  | 0 | 0 | 0 |  | 0
    Period 2: Withdrawal vs Continued Tx: Unknown or Not Reported |  | 0 | 0 | 0 |  | 0
    Period 2: Open-Label Retreatment: number analyzed (Participants) | 0 | 0 | 0 | 0 | 63 | 63
    Period 2: Open-Label Retreatment: American Indian or Alaska Native |  |  |  |  | 0 | 0
    Period 2: Open-Label Retreatment: Asian |  |  |  |  | 0 | 0
    Period 2: Open-Label Retreatment: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0
    Period 2: Open-Label Retreatment: Black or African American |  |  |  |  | 0 | 0
    Period 2: Open-Label Retreatment: White |  |  |  |  | 63 | 63
    Period 2: Open-Label Retreatment: More than one race |  |  |  |  | 0 | 0
    Period 2: Open-Label Retreatment: Unknown or Not Reported |  |  |  |  | 0 | 0
C-Reactive Protein (CRP) Category at Enrollment [Count of Participants; unit: Participants] — Population: The first row represents Period 1, the second row represents the double-blind portion of Period 2, and the third row represents open-label retreatment in Period 2
  Participants
    Period 1: Open-Label Run-In: number analyzed (Participants) | 323 | 0 | 0 | 0 | 0 | 323
    Period 1: Open-Label Run-In: > 6 mg/L | 196 |  |  |  |  | 196
    Period 1: Open-Label Run-In: ≤ 6 mg/L | 127 |  |  |  |  | 127
    Period 2: Withdrawal vs Continued Tx: number analyzed (Participants) | 0 | 63 | 64 | 62 | 0 | 189
    Period 2: Withdrawal vs Continued Tx: > 6 mg/L |  | 40 | 40 | 39 |  | 119
    Period 2: Withdrawal vs Continued Tx: ≤ 6 mg/L |  | 23 | 24 | 23 |  | 70
    Period 2: Open-Label Retreatment: number analyzed (Participants) | 0 | 0 | 0 | 0 | 63 | 63
    Period 2: Open-Label Retreatment: > 6 mg/L |  |  |  |  | 38 | 38
    Period 2: Open-Label Retreatment: ≤ 6 mg/L |  |  |  |  | 25 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without a Disease Activity Flare During Period 2
Description: Disease flare is defined as an Ankylosing Spondylitis Disease Activity Score (ASDAS) at two consecutive visits that both show either absolute score ≥2.1 or a post-withdrawal increase of ≥1.1 relative to baseline prior to the first dose of double-blind treatment in Period 2. The ASDAS is a composite index assessing disease activity in axial spondyloarthropathies that consists of 4 self-assessed parameters and 1 laboratory parameter. The self-assessed parameters of back pain, duration of morning stiffness, Patient Global Disease Assessment (PGDn), and peripheral pain/swelling are individually scored on a numeric scale of 0 to 10, with 0 being low activity/impact and 10 being high activity/impact. The self-assessed criteria and the laboratory value of CRP are combined to provide the total ASDAS score, which has a lower limit of 0.6 and no defined upper limit. A higher score indicates greater disease activity.
Time Frame: Up to 12 months
Population: The analysis population consists of all participants who attained inactive disease in Period 1, were randomized in Period 2, and received at least one dose of double-blind study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 84.1 | 68.3 | 33.9
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; p < 0.001, Miettinen and Nurminen; Derived based on the stratified Miettinen and Nurminen method with CRP level (>6 mg/L or ≤ 6 mg/L) as a stratification factor; Difference in percentage = 50.2, 95% CI 2-sided [34.1 to 63.6]
Statistical Analysis 2: Comparison: Golimumab Q2M (Reduced Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; p < 0.001, Meittinen and Nurminen; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 34.4, 95% CI 2-sided [17.0 to 49.7]

2. Secondary Outcome: Percentage of Participants With a Flare Who Show a Clinical Response Within 3 Months of Open-Label Golimumab Retreatment
Description: Clinical response is defined as Bath Ankylosing Spondylitis Disease Assessment Index (BASDAI) score improvement of ≥2.0 or ≥50% improvement within 3 months of the start of retreatment, relative to the mean of the two consecutive BASDAI scores that defined the flare. Sustained clinical response refers to participants who attained clinical response and maintained BASDAI criteria throughout the 3-month retreatment period. Response data was collected throughout Period 2 (12 months) and censored to include only the first 3 months after retreatment for a disease flare. The BASDAI is a summary of 6 participant-assessed measures rated on scales of 0 (none) to 10 (very severe): fatigue, spinal pain, joint pain/swelling, tenderness, morning stiffness, and duration of morning stiffness [0 (zero) to 10 (2 or more hours)]. The BASDAI score is the mean of responses to the 6 questions with a minimum of 0 and a maximum of 10. A higher score indicates greater disease activity.
Time Frame: Up to 3 months following start of retreatment
Population: The analysis population consists of all participants who attained inactive disease in Period 1, were randomized to the reduced-treatment regimen or placebo in Period 2, received at least one dose of double-blind study intervention, and experienced a disease flare during Period 2. Per protocol, participants randomized to the Full Treatment Regimen were not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Retreatment
Number analyzed (Participants) | 53
Percentage of participants
  Within 1 month of retreatment | 90.6 [79.3 to 96.9]
  Within 2 months of retreatment | 96.2 [87.0 to 99.5]
  Within 3 months of retreatment | 96.2 [87.0 to 99.5]
  Sustained clinical response | 71.7 [57.7 to 83.2]

3. Secondary Outcome: Time to First Disease Flare
Description: The Kaplan-Meier analysis of time to first "flare" in Period 2 is represented by the percentage of participants who experienced a disease flare relative to baseline prior to the first dose of double-blind treatment in Period 2. Disease flare is defined as ASDAS at two consecutive visits that both show either absolute score ≥2.1 or a post-withdrawal increase of ≥1.1.
Time Frame: Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants
  Month 3 | 14.3 | 7.9 | 41.9
  Month 6 | 14.3 | 17.5 | 58.1
  Month 9 | 14.3 | 20.6 | 61.3
  Month 12 | 15.9 | 23.8 | 61.3

4. Secondary Outcome: Percentage of Participants Achieving ASAS20 (Assessment in SpondyloArthritis International Society) Response (Double-blind Treatment)
Description: ASAS20 is a 20% improvement in response (per the Assessment in Ankylosing Spondylitis International Working Group) defined as meeting 2 criteria: 1) An improvement of ≥20% from Baseline and an absolute improvement from Baseline of ≥1.0 in at least 3 of 4 domains, and 2) Absence of deterioration from Baseline (defined as a ≥20% worsening and an absolute worsening of ≥1.0) in the potential remaining domain. Baseline for ASAS20 analysis is defined as the last ASAS score prior to the first dose of double-blind treatment in Period 2. The ASAS consists of 4 domains: the Patient Global Disease Assessment (PGDn), total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and morning stiffness (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 10-point numeric scale from 0=no disease symptoms/impact to 10=extreme disease symptoms/impact, with a higher score indicating more severe impairment.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 9.5 | 3.2 | 0.0
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 9.5, 95% CI 2-sided [3.3 to 19.4] — Derived based on the stratified Miettinen and Nurminen method with CRP level (>6 mg/L or ≤ 6 mg/L) as a stratification factor
Statistical Analysis 2: Comparison: Golimumab Q2M (Reduced Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 3.2, 95% CI 2-sided [-2.8 to 10.9] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving ASAS20 Response (Open-label Retreatment)
Description: ASAS20 is a 20% improvement in response (per the Assessment in Ankylosing Spondylitis International Working Group) defined as meeting 2 criteria: 1) An improvement of ≥20% from Baseline and an absolute improvement from Baseline of ≥1.0 in at least 3 of 4 domains, and 2) Absence of deterioration from Baseline (defined as a ≥20% worsening and an absolute worsening of ≥1.0) in the potential remaining domain. Baseline for ASAS20 analysis is defined as the last ASAS score prior to the first dose of open-label retreatment in Period 2. The ASAS consists of 4 domains: the Patient Global Disease Assessment (PGDn), total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and morning stiffness (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 10-point numeric scale from 0=no disease symptoms/impact to 10=extreme disease symptoms/impact, with a higher score indicating more severe impairment.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Retreatment
Number analyzed (Participants) | 53
Percentage of participants | 94.3 [84.3 to 98.8]

6. Secondary Outcome: Percentage of Participants Achieving ASAS40 Response (Double-blind Treatment)
Description: ASAS40 is a 40% improvement in response (per the Assessment in Ankylosing Spondylitis International Working Group) defined as meeting 2 criteria: 1) An improvement of ≥40% from Baseline and an absolute improvement from Baseline of ≥2.0 in at least 3 of 4 domains, and 2) No deterioration from Baseline in the potential remaining domain. Baseline for ASAS40 analysis is defined as the last ASAS score prior to the first dose of double-blind treatment in Period 2. The ASAS consists of 4 domains: the Patient Global Disease Assessment (PGDn), total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and morning stiffness (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 10-point numeric scale from 0=no disease symptoms/impact to 10=extreme disease symptoms/impact, with a higher score indicating more severe impairment.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 0.0, 95% CI 2-sided [-5.9 to 5.8] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Q2M (Reduced Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 0.0, 95% CI 2-sided [-5.9 to 5.8] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Percentage of Participants Achieving ASAS40 Response (Open-label Retreatment)
Description: ASAS40 is a 40% improvement in response (per the Assessment in Ankylosing Spondylitis International Working Group) defined as meeting 2 criteria: 1) An improvement of ≥40% from Baseline and an absolute improvement from Baseline of ≥2.0 in at least 3 of 4 domains, and 2) No deterioration from Baseline in the potential remaining domain. Baseline for ASAS40 analysis is defined as the last ASAS score prior to the first dose of open-label retreatment in Period 2. The ASAS consists of 4 domains: the Patient Global Disease Assessment (PGDn), total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and morning stiffness (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 10-point numeric scale from 0=no disease symptoms/impact to 10=extreme disease symptoms/impact, with a higher score indicating more severe impairment.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Retreatment
Number analyzed (Participants) | 53
Percentage of participants | 90.6 [79.3 to 96.9]

8. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission (Double-blind Treatment)
Description: ASAS partial remission is defined as a score of ≤2 in all 4 ASAS domains. Baseline for this analysis is defined as the ASAS score prior to the first dose of double-blind treatment in Period 2. The ASAS consists of 4 domains: Patient Global Disease Assessment (PGDn), total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and morning stiffness (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 10-point numeric scale from 0=no disease symptoms/impact to 10=extreme disease symptoms/impact, with a higher score indicating more severe impairment.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 85.7 | 85.7 | 71.0
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 14.7, 95% CI 2-sided [0.2 to 29.0] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Q2M (Reduced Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 14.7, 95% CI 2-sided [0.2 to 29.1] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission (Open-label Retreatment)
Description: ASAS partial remission is defined as a score of ≤2 in all 4 ASAS domains. Baseline for this analysis is defined as the ASAS score prior to the first dose of open-label retreatment in Period 2. The ASAS consists of 4 domains: Patient Global Disease Assessment (PGDn), total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and morning stiffness (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 10-point numeric scale from 0=no disease symptoms/impact to 10=extreme disease symptoms/impact, with a higher score indicating more severe impairment.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Retreatment
Number analyzed (Participants) | 53
Percentage of participants | 92.5 [81.8 to 97.9]

10. Secondary Outcome: Percentage of Participants Achieving BASDAI50 Response (Double-blind Treatment)
Description: BASDAI50 is defined as ≥50% improvement from baseline in the Bath Ankylosing Spondylitis Disease Assessment Index (BASDAI) score. Baseline for BASDAI50 analysis is defined as the last BASDAI score prior to the first dose of double-blind treatment in Period 2. The BASDAI is a summary of 6 participant-assessed measures rated on scales of 0 (none) to 10 (very severe): fatigue, spinal pain, joint pain/swelling, tenderness, morning stiffness, and duration of morning stiffness [0 (zero) to 10 (2 or more hours)]. The BASDAI score is the mean of responses to the 6 questions with a minimum of 0 and a maximum of 10. A higher score indicates greater disease activity.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 49.2 | 30.2 | 24.2
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 24.9, 95% CI 2-sided [8.5 to 40.3] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Q2M (Reduced Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 5.9, 95% CI 2-sided [-9.9 to 21.3] — [estimate comment as in outcome 4, analysis 1]

11. Secondary Outcome: Percentage of Participants Achieving BASDAI50 Response (Open-label Retreatment)
Description: BASDAI50 is defined as ≥50% improvement from baseline in the Bath Ankylosing Spondylitis Disease Assessment Index (BASDAI) score. Baseline for BASDAI50 analysis is defined as the last BASDAI score prior to the first dose of open-label retreatment in Period 2. The BASDAI is a summary of 6 participant-assessed measures rated on scales of 0 (none) to 10 (very severe): fatigue, spinal pain, joint pain/swelling, tenderness, morning stiffness, and duration of morning stiffness [0 (zero) to 10 (2 or more hours)]. The BASDAI score is the mean of responses to the 6 questions with a minimum of 0 and a maximum of 10. A higher score indicates greater disease activity.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Retreatment
Number analyzed (Participants) | 53
Percentage of participants | 98.1 [89.9 to 100.0]

12. Secondary Outcome: Percentage of Participants Achieving Inactive Disease Status (Double-Blind Treatment)
Description: Inactive disease status is defined as an ASDAS score <1.3. The ASDAS is a composite index assessing disease activity in axial spondyloarthropathies that consists of 4 self-assessed parameters and 1 laboratory parameter. The self-assessed parameters of back pain, duration of morning stiffness, Patient Global Disease Assessment (PGDn), and peripheral pain/swelling are individually scored on a numeric scale of 0 to 10, with 0 being low activity/impact and 10 being high activity/impact. The self-assessed criteria and the laboratory value of CRP are combined to provide the total ASDAS score, which has a lower limit of 0.6 and no defined upper limit. A higher score indicates greater disease activity.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen)
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 85.7 | 84.1 | 61.3
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 24.4, 95% CI 2-sided [9.1 to 39.0] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Q2M (Reduced Treatment Regimen) vs Placebo (Treatment Withdrawal Regimen); Test type: Superiority; Difference in percentage = 22.8, 95% CI 2-sided [7.3 to 37.7] — [estimate comment as in outcome 4, analysis 1]

13. Secondary Outcome: Percentage of Participants Achieving Inactive Disease Status (Open-label Retreatment)
Description: as for outcome 12
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Open-Label Retreatment
Number analyzed (Participants) | 53
Percentage of participants | 90.6 [79.3 to 96.9]

14. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE) in Period 2
Description: This endpoint evaluated the safety and tolerability of withdrawing from or continuing treatment with golimumab in Period 2. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of study treatment, is also an AE. The analysis includes AEs that occurred through 90 days after the last dose of study treatment.
Time Frame: Up to approximately 15 months
Population: The analysis population consists of all participants who received at least one dose of study intervention in Period 2.
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment
Number analyzed (Participants) | 63 | 64 | 62 | 63
Percentage of participants | 46.0 | 46.9 | 32.3 | 41.3

15. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE in Period 2
Description: This endpoint evaluated the safety and tolerability of withdrawing from or continuing treatment with golimumab in Period 2. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of study treatment, is also an AE.
Time Frame: Up to approximately 12 months
Population: The analysis population consists of all participants who received at least one dose of study intervention in Period 2.
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment
Number analyzed (Participants) | 63 | 64 | 62 | 63
Percentage of participants | 0.0 | 4.7 | 1.6 | 0.0

16. Other Pre Specified Outcome: Percentage of Participants Without a Disease Activity Flare During Period 2 (Full Treatment Regimen Versus Withdrawal Regimens)
Description: as for outcome 1
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Golimumab QM (Full Treatment Regimen): Participants were treated with double-blinded SC injections of 50 mg golimumab QM for up to 12 months. Participants with a body weight greater than 100 kg who had received 100 mg injections of golimumab in Period 1 continued to receive this dosage for the duration of the study.
- Golimumab Q2M and Placebo (Withdrawal Regimens): Participants were treated with double-blinded SC injections of 50 mg golimumab Q2M alternating with matching placebo to golimumab every other month or with placebo for up to 12 months. Participants with a body weight greater than 100 kg who had received 100 mg injections of golimumab in Period 1 continued to receive this dosage for the duration of the study.
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M and Placebo (Withdrawal Regimens)
Number analyzed (Participants) | 63 | 125
Percentage of participants | 84.1 | 51.2
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Golimumab Q2M and Placebo (Withdrawal Regimens); Test type: Superiority; p < 0.001, Miettinen and Nurminen; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 32.9, 95% CI 2-sided [19.2 to 44.5]

17. Other Pre Specified Outcome: Percentage of Participants Without a Disease Activity Flare During Period 2 (Full Treatment Regimen Versus Reduced Treatment Regimen)
Description: as for outcome 1
Time Frame: Up to 12 months
Population: The analysis population consists of all participants who attained inactive disease in Period 1, were randomized to receive golimumab in Period 2, and received at least one dose of double-blind study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen)
Number analyzed (Participants) | 63 | 63
Percentage of participants | 84.1 | 68.3
Statistical Analysis 1: Comparison: Golimumab QM (Full Treatment Regimen) vs Golimumab Q2M (Reduced Treatment Regimen); Test type: Superiority; p = 0.037, Miettinen and Nurminen; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 15.9, 95% CI 2-sided [0.9 to 30.5]

ADVERSE EVENTS:
Time Frame: Up to 10 months in Period 1 (Open-Label Run-in) and up to 15 months in Period 2 (Withdrawal vs Continued Treatment) for a total of up to 25 months.
Description: The safety analysis population includes all participants who received at least one dose of study intervention.
Arm/Group | Open-Label Run-In Golimumab QM | Golimumab QM (Full Treatment Regimen) | Golimumab Q2M (Reduced Treatment Regimen) | Placebo (Treatment Withdrawal Regimen) | Open-Label Retreatment
All-Cause Mortality (participants affected / at risk) | 0/323 | 0/63 | 0/64 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 7/323 | 1/63 | 1/64 | 1/62 | 0/63
Other Adverse Events (participants affected / at risk) | 79/323 | 13/63 | 17/64 | 11/62 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Run-In Golimumab QM (N=323) | Golimumab QM (Full Treatment Regimen) (N=63) | Golimumab Q2M (Reduced Treatment Regimen) (N=64) | Placebo (Treatment Withdrawal Regimen) (N=62) | Open-Label Retreatment (N=63)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Run-In Golimumab QM (N=323) | Golimumab QM (Full Treatment Regimen) (N=63) | Golimumab Q2M (Reduced Treatment Regimen) (N=64) | Placebo (Treatment Withdrawal Regimen) (N=62) | Open-Label Retreatment (N=63)
Nasopharyngitis (Infections and infestations) | 36 (39) | 6 (7) | 6 (6) | 3 (4) | 4 (4)
Pharyngitis (Infections and infestations) | 12 (14) | 2 (2) | 6 (9) | 3 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (24) | 2 (5) | 3 (3) | 2 (3) | 5 (5)
Headache (Nervous system disorders) | 24 (39) | 4 (8) | 2 (3) | 4 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03253796/Prot_SAP_000.pdf